CLINICAL TRIAL: NCT04223271
Title: Noninvasive Home Assessment of Cardiac Filling Pressure to Identify Heart Failure Patients at High Risk for Readmission
Brief Title: Heart Failure Event Advance Detection Trial
Acronym: HEADstart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vixiar Medical, Inc. (Industry)
Collaborators: Johns Hopkins University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PROT000035; 1R42HL136162 (NIH)
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-03

CONDITIONS: Congestive Heart Failure; Heart Failure; Decompensated Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Acutely Decompensated Heart Failure Patients: Patients who are admitted with acutely decompensated heart failure and are receiving intravenous diuretics will be recruited to undergo testing. Testing with the Indicor device will occur every day during hospitalization, and twice a day for up to 30 days after discharge.
  Interventions: Diagnostic Test: Indicor

INTERVENTIONS:
Diagnostic Test: Indicor — Handheld device with attached PPG sensor that is paired with a tablet to estimate left ventricular end diastolic pressure. Subjects will blow into the device in order to perform a standardized Valsalva maneuver for 10 seconds. The index finger will be resting in the PPG sensor during the test. Each test requires three efforts, with 45 seconds rest between efforts.

SUMMARY:
Patients who are admitted with acutely decompensated heart failure and are receiving intravenous diuretics will be recruited to undergo testing using the Indicor Device. Participants will be tested daily while hospitalized and then on the day of discharge during which time they will be trained how to operate the device. Once discharged, patients will perform one test in the morning, and one test in the evening for up to 30 days.

DETAILED DESCRIPTION:
The study will follow the design of a prospective observational cohort study. Patients who are admitted with acutely decompensated heart failure and are receiving intravenous diuretics will be recruited to undergo testing with the Indicor Device for estimating left ventricular end diastolic pressure (LVEDP). Trends in estimated LVEDP will be assessed after thirty days at home to identify trends that coincided with heart failure events.

The Indicor is a noninvasive device that assesses cardiac filling pressure based on the long understood phenomenon that performing a Valsalva maneuver induces changes in pulse pressure that reflect cardiac filling pressure.Testing with the Indicor consists of blowing into the device while performing a Valsalva Maneuver for 10 seconds, and the index finger will be placed inside a PPG sensor during the test. Each test consists of three recorded efforts with 45 seconds rest between efforts.

Participants will be tested daily while hospitalized and then on the day of discharge during which time they will be trained how to operate the device. In order to proceed with home use, they will need to demonstrate the ability to properly operate the device and complete testing without assistance. Demographic and clinical data will also be collected including laboratories, comorbidities, and heart failure etiology. Once a subject demonstrates proper operation an Indicor will be provided to them for use at home for the study duration. Once the subjects are home, they will be asked to perform the test each morning and each evening.

In the AM, subjects will be asked to weigh themselves upon awakening after using the restroom, and will be asked to perform the device test afterward. Subjects will be asked six simple, standardized symptom-related questions:

1. Have you felt more short of breath during the last day?
2. Have you noticed more swelling in the last day?
3. Did you wake up short of breath last night?
4. Did you sleep in a chair, or prop up with pillows more than usual last night?
5. Have you had any lightheadedness or dizziness in the last day?
6. Enter morning weight.

No recorded data will be analyzed for the duration of the subject's participation, since this is purely an observational study. It will be stressed to the participant that, as always, they would need to report to their provider any worsening symptoms or change in weight as instructed by the discharge team or outpatient provider.

For each subject enrolled, 1 test twice a day will be obtained for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Johns Hopkins Hospital, or Johns Hopkins Bayview Medical Center with acutely decompensated heart failure (HFrEF or HFpEF)
* Requires IV diuresis

Exclusion Criteria:

* Acute coronary syndrome (type 1 myocardial infarction)
* Terminal non-cardiac illness (that can affect short term prognosis)
* Operative cardiac procedure during admission (bypass, valve, transplant, LVAD)
* End-stage renal disease on dialysis
* Pregnant women (as verbally indicated by patients being approached for recruitment, or through clinically indicated pregnancy tests ordered by the patient's clinicians)
* History of paradoxical emboli
* Hypertrophic obstructive cardiomyopathy
* Known intracardiac shunt
* Known severe aortic valve stenosis
* Known severe mitral valve stenosis
* Myocardial infarction within one week of intended Indicor testing
* Uncontrolled hypertension (systolic BP >160mmHg or diastolic BP> 100mmHg)
* Hypotension (systolic BP <90mmHg)
* Symptomatic bradycardia
* Known cholesterol emboli
* Poor left ventricular function with left ventricular thrombus
* Unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient admitted to Johns Hopkins Hospital, or Johns Hopkins Bayview Medical Center with acutely decompensated heart failure (HFrEF or HFpEF) that does not meet any of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Association between change in estimated LVEDP and the occurrence of heart failure events. | 30 days post discharge
  Twice daily, non-invasive measures to estimate LVEDP (mmHg) will be retrospectively assessed to determine if changes or trends in estimated LVEDP were associated with, and therefore predictive of, 30-day readmission, mortality or need for intravenous diuretics in heart failure patients.

CONTACTS AND LOCATIONS:
Overall Officials: Harry A Silber, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No